CLINICAL TRIAL: NCT05238467
Title: Long Term Immunological Responses of COVID-19 Vaccination in Cancer Patients on Chemotherapy: a Pilot Study
Brief Title: Immunological Responses of COVID-19 Vaccination
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Alberto J. Montero, Professor of Medicine, University Hospitals Cleveland Medical Center
Other Study IDs: STUDY20210455
Record Dates: First submitted 2022-02-10; First posted 2022-02-14 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Cancer; Chemotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- A: Group A will consist of 50 participants with a diagnosis of one of the following cancers: breast, colorectal, or prostate cancers who received myelosuppressive cytotoxic chemotherapy at the time of COVID vaccination, or who received chemotherapy within 30 days prior to the initial or booster vaccination, or who started on chemotherapy within 30 days after the initial or booster COVID vaccination. Cytotoxic chemotherapy can be given either in the neoadjuvant/adjuvant setting or metastatic setting.
  Interventions: Other: COVID antibody titers in the blood
- B: Group B will consist of 25 participants with a diagnosis of breast, colorectal, or prostate cancers who are on non-myelosuppressive treatment including endocrine therapy, tyrosine kinase inhibitor or anti-HER 2 therapy.
  Interventions: Other: COVID antibody titers in the blood
- C: Group C will consist of 25 age matched adult participants with no prior history of cancer or prior history of non-metastatic solid cancer invasive cancer treated with a curative intent, without evidence of disease recurrence, and >12 months from completion of chemotherapy or radiation.
  Interventions: Other: COVID antibody titers in the blood

INTERVENTIONS:
Other: COVID antibody titers in the blood — COVID antibody titers will be quantitatively assessed at baseline, 8 weeks and approximately 6, 9, and 12 months from date of study enrollment. Titers will be compared to levels in 25 age matched adult participants with no prior history of cancer or prior history of non-metastatic solid cancer invasive cancer treated with a curative intent,.and in 25 age matched cancer participants who are on non-immunosuppressive treatments as defined below.

SUMMARY:
Cancer patients with COVID-19 have a 30% higher mortality rate compared to the general population and are considered a high-risk group by the American Association for Cancer Research that should be given "high priority" during COVID-19 vaccine administration. Although studies have suggested that vaccination during active treatment with chemo and/or radiation therapy provides suboptimal antibody response, the studies were underpowered and heterogeneous thus putting this conclusion into question. We need data in cancer patients on immunosuppressive chemotherapy at the time of COVID vaccination to understand how immune responses compare to healthy controls and cancer patients not on immunosuppressive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following inclusion criteria to be eligible for enrollment:

  1. Willing and able to provide written informed consent for the trial.
  2. Male or female participants >18 years of age on the day of signing informed consent.
  3. a. Participants (>18 years) with gastrointestinal (gastroesophageal, pancreatic, small bowel, colon, anal) solid tumors, breast, or prostate cancers who received myelosuppressive chemotherapy within 60 days prior to initial or booster COVID vaccination, or who started on chemotherapy within 60 days after the initial or booster COVID vaccination; or b. Adult participants (>18 years) not receiving chemotherapy at the time of initial or booster COVID vaccination, but who were on non-immunosuppressive treatments (endocrine therapy, treatment with tyrosine kinase inhibitor or antiHER-2 therapy); or c. Adult participants > 18 years either: (i) with no history of cancer or (ii) prior history of non-metastatic solid cancer invasive cancer treated with a curative intent, without evidence of disease recurrence, and >12 months from completion of chemotherapy or radiation.
  4. a. Participants in groups A and B who have a planned COVID vaccination within the next 90 days of study enrollment with any FDA approved vaccine, or previous COVID vaccination within 90 days from study enrollment are eligible provided they meet all other above eligibility criteria; or b. Participants in group C who have planned COVID vaccination within the next 90 days of study enrollment with any FDA approved vaccine; or previous COVID vaccination within six months from study enrollment are eligible provided they meet all other above eligibility criteria

Exclusion Criteria:

* Participants will be considered ineligible for enrollment with the following criteria:

  1. Participants currently on immunotherapy
  2. Participants with documented COVID 19 infection within < 6 months from study enrollment
  3. Prior history of autoimmune disorder and are currently on immunosuppressive therapy or have received immunosuppressive therapy within the last 6-12 months prior to enrollment
  4. No planned and no prior COVID vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group A will consist of 50 participants with a diagnosis of one of the following cancers: breast, colorectal, or prostate cancers who received myelosuppressive cytotoxic chemotherapy at the time of COVID vaccination, or who received chemotherapy within 30 days prior to the initial or booster vaccination, or who started on chemotherapy within 30 days after the initial or booster COVID vaccination. Group B will consist of 25 participants with a diagnosis of breast, colorectal, or prostate cancers who are on non-myelosuppressive treatment including endocrine therapy, tyrosine kinase inhibitor or anti-HER 2 therapy. Group C will consist of 25 age matched adult participants with no prior history of cancer or prior history of non-metastatic solid cancer invasive cancer treated with a curative intent, without evidence of disease recurrence, and >12 months from completion of chemotherapy or radiation.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Seroprotection rate | 05/2021-12/31/2022
  had an antibody titer protective (1:40) at any point in testing

SECONDARY OUTCOMES:
Seroconversion rate | 05/2021-12/31/2022
  the proportion of participants who had an antibody titer fourfold increase in their antibody titer to 1:40 or greater after vaccination over baseline

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Desai A, Sachdeva S, Parekh T, Desai R. COVID-19 and Cancer: Lessons From a Pooled Meta-Analysis. JCO Glob Oncol. 2020 Apr;6:557-559. doi: 10.1200/GO.20.00097. No abstract available. PMID 32250659
- [Background] Desai A, Gupta R, Advani S, Ouellette L, Kuderer NM, Lyman GH, Li A. Mortality in hospitalized patients with cancer and coronavirus disease 2019: A systematic review and meta-analysis of cohort studies. Cancer. 2021 May 1;127(9):1459-1468. doi: 10.1002/cncr.33386. Epub 2020 Dec 30. PMID 33378122
- [Background] Kuderer NM, Choueiri TK, Shah DP, Shyr Y, Rubinstein SM, Rivera DR, Shete S, Hsu CY, Desai A, de Lima Lopes G Jr, Grivas P, Painter CA, Peters S, Thompson MA, Bakouny Z, Batist G, Bekaii-Saab T, Bilen MA, Bouganim N, Larroya MB, Castellano D, Del Prete SA, Doroshow DB, Egan PC, Elkrief A, Farmakiotis D, Flora D, Galsky MD, Glover MJ, Griffiths EA, Gulati AP, Gupta S, Hafez N, Halfdanarson TR, Hawley JE, Hsu E, Kasi A, Khaki AR, Lemmon CA, Lewis C, Logan B, Masters T, McKay RR, Mesa RA, Morgans AK, Mulcahy MF, Panagiotou OA, Peddi P, Pennell NA, Reynolds K, Rosen LR, Rosovsky R, Salazar M, Schmidt A, Shah SA, Shaya JA, Steinharter J, Stockerl-Goldstein KE, Subbiah S, Vinh DC, Wehbe FH, Weissmann LB, Wu JT, Wulff-Burchfield E, Xie Z, Yeh A, Yu PP, Zhou AY, Zubiri L, Mishra S, Lyman GH, Rini BI, Warner JL; COVID-19 and Cancer Consortium. Clinical impact of COVID-19 on patients with cancer (CCC19): a cohort study. Lancet. 2020 Jun 20;395(10241):1907-1918. doi: 10.1016/S0140-6736(20)31187-9. Epub 2020 May 28. PMID 32473681
- [Background] Ribas A, Sengupta R, Locke T, Zaidi SK, Campbell KM, Carethers JM, Jaffee EM, Wherry EJ, Soria JC, D'Souza G; AACR COVID-19 and Cancer Task Force. Priority COVID-19 Vaccination for Patients with Cancer while Vaccine Supply Is Limited. Cancer Discov. 2021 Feb;11(2):233-236. doi: 10.1158/2159-8290.CD-20-1817. Epub 2020 Dec 19. PMID 33355178
- [Background] Ljungman P. Vaccination of immunocompromised patients. Clin Microbiol Infect. 2012 Oct;18 Suppl 5:93-9. doi: 10.1111/j.1469-0691.2012.03971.x. PMID 23051059